CLINICAL TRIAL: NCT06358976
Title: The Effectiveness of Anti-spastic Splint With Added Focal Muscle Vibration (FMV) in Decreasing Hand Spasticity and Improving Hand Functionality Among Individuals With Chronic Stroke: a Pilot Randomized Control Trial
Brief Title: Anti-Spastic Splint With Focal Muscle Vibration for Stroke Hand Spasticity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arab American University (Palestine) (Other)
Responsible Party: Principal Investigator, Amer Jaroshy, Principal Investigator, Arab American University (Palestine)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: Spasticity splint and FMV
Record Dates: First submitted 2024-04-06; First posted 2024-04-11 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Spasticity as Sequela of Stroke
Keywords: Stroke; Spasticity; Vibration; Splint; Upper limb
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Vibration

STUDY DESIGN:
Intervention Model Description: The interventional study model for this clinical study is a pilot randomized controlled trial. Participants will be randomly assigned to one of three arms: Group A (vibrating splint intervention), Group B (standard splint intervention), or Group C (control group receiving no splint intervention). This model allows for the comparison of different interventions and the evaluation of their effectiveness in improving hand function and reducing spasticity after stroke. Randomization helps ensure that each group is comparable in terms of baseline characteristics, minimizing bias and increasing the validity of the study results.
Who Masked: Investigator
Masking Description: In this clinical trial, due to the nature of the interventions, it may not be possible to mask or blind the participants or therapists to the treatment received. However, efforts will be made to blind the outcome assessors who will be responsible for evaluating the participants' hand function, spasticity, and other outcome measures. Blinding the outcome assessors helps minimize potential bias and ensures the objective assessment of the intervention's effectiveness. By keeping the assessors unaware of the participants' group allocations, the integrity and reliability of the study findings can be enhanced.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vibration plus anti-spastic hand splint Arm (Experimental): In this clinical trial, vibration stimulation will be applied to the spastic hand antagonistic muscles using a specific device consisting of a volar anti-spastic hand splint and the arm vibrator. The volar anti-spastic hand splint will be custom-made for each participant at the prosthetic and orthotic clinic, following a standardized protocol. The arm vibrator, designed to fit the arm, will deliver the required vibration parameters. The intervention protocol involves a 30-minute vibration session administered three times weekly for four weeks, accompanied by daily utilization of the custom-made splint for 30 minutes each day.
  Interventions: Other: Vibration plus anti-spastic hand splint
- Anti-spastic hand splint Arm (Active Comparator): In the anti-spastic hand splint arm , participants will be provided with an anti-spastic splint without vibration. Both vibration plus anti-spastic hand splint arm and anti-spastic hand splint arm will adhere to the same splint standard regime and recommendations, which outlines the specific positioning for the splint.
  Interventions: Other: Anti-spastic hand splint
- Vibration Arm (Active Comparator): In vibration arm , participants will be provided with arm vibrator held in place by appropriate padded harness. A Standardized study protocol will be used each time with no splint.
  Interventions: Other: Vibration

INTERVENTIONS:
Other: Vibration plus anti-spastic hand splint — vibration stimulation will be applied to the spastic hand antagonistic muscles using a volar anti-spastic hand splint and the Myovolt Arm vibrator.
  Arms: Vibration plus anti-spastic hand splint Arm
Other: Anti-spastic hand splint — the use of anti-spastic hand splint alone.
  Arms: Anti-spastic hand splint Arm
Other: Vibration — The use of hand vibrator alone
  Arms: Vibration Arm

SUMMARY:
Title: The Effect of Vibrating Splint on Hand Function After Stroke

Summary:

This study aims to investigate the effectiveness of a vibrating splint in improving hand function and reducing spasticity among individuals who have experienced a stroke. Stroke is a major global health issue, often resulting in long-term disability and impairments in the upper limbs. Spasticity, a common complication of stroke, causes stiffness and involuntary muscle contractions, leading to difficulties in performing daily activities.

Current treatment options for spasticity include medications and physical therapy techniques. However, these approaches may have limitations in terms of effectiveness and duration of benefits. Therefore, non-pharmacological interventions are being explored to enhance rehabilitation outcomes.

The hypothesis of this study is that the use of a vibrating splint, which applies mechanical vibrations to the hand muscles, will decrease spasticity and improve hand functionality in individuals with chronic stroke. The vibrations from the splint stimulate the sensory receptors in the skin and muscles, leading to muscle relaxation and improved motor control.

The study will be conducted as a pilot randomized controlled trial, involving participants who meet specific eligibility criteria. The participants will be divided into three arms, with each arm receiving a different intervention. Outcome measures, including assessments of spasticity, range of motion, pain levels, and functional abilities, will be collected before and after the intervention period.

The findings from this study will contribute to the understanding of non-pharmacological approaches in managing spasticity and improving hand function after stroke. If the vibrating splint proves to be effective, it could offer a safe and accessible option for stroke survivors to enhance their recovery and regain independence in daily activities.

This research is essential as it addresses the need for more effective interventions for spasticity management and hand rehabilitation after stroke. By providing valuable insights into the potential benefits of the vibrating splint, this study has the potential to improve the quality of life for individuals who have experienced a stroke and empower them to regain control over their hand movements.

DETAILED DESCRIPTION:
This pilot randomized controlled trial (RCT) aims to assess the clinical effectiveness and efficacy of adding focal muscle vibration (FMV) to anti-spastic splint therapy for individuals with spasticity following a stroke. The study involves multiple centers in the Jenin area of Palestine, utilizing outpatient rehabilitation centers to recruit participants who have chronic spasticity post-stroke.

Study Objectives and Questions:

Determine whether adding FMV to anti-spastic splint therapy provides additional benefit for individuals with spasticity after a stroke.

Compare the outcomes of anti-spastic splint therapy, FMV therapy, and a combination of both interventions in individuals with post-stroke spasticity.

Explore participant perceptions regarding the effectiveness, acceptability, and adherence to the interventions.

Study Design and Procedures:

The study is a pilot, multi-center RCT with a single evaluator (evaluator-blind) approach to avoid bias.

Forty-eight participants will be randomly assigned to one of three groups: Arm 1 (anti-spastic splint and FMV), Arm 2 (FMV only), or Arm 3 (anti-spastic splint only).

Interventions will be delivered by trained rehabilitation specialists, including occupational and physical therapists.

Standardized intervention protocols will guide the delivery of FMV and anti-spastic splint therapy for a period of four weeks.

Participant Recruitment:

Participants with chronic post-stroke spasticity are recruited from multiple rehabilitation centers and screened based on specific inclusion and exclusion criteria.

Convenience sampling is used to enroll participants from available populations in the participating centers.

Data Collection and Management:

Baseline and post-treatment evaluations include measurements of spasticity, hand functionality, range of motion, and pain level.

Qualitative interviews will explore participants' experiences with the interventions and their perceptions of the treatments' effectiveness.

Data will be securely stored and anonymized to protect participants' privacy.

Statistical Analysis Plan:

Linear Mixed-Effects Models (LMEM) will be used to assess treatment effects, adjusting for correlation over time within participants.

The safety analysis will involve documenting and summarizing adverse events (AEs) across treatment groups.

The study aims to provide preliminary data on treatment effects and inform the design of future larger RCTs.

ELIGIBILITY:
Inclusion Criteria:

* Individuals affected by chronic (more than one year) spastic ischemic or hemorrhagic stroke
* Aged above 18 years old
* Medically stable (has no cardiovascular event in the last 12 months)
* A score of 1-4 on modified Ashworth scale.

Exclusion Criteria:

* Cardiovascular event in the past 12 months
* Received anti-spastic injections drugs into the affected hand in the last 6 months
* A score of less than 21 on Rowland Universal Dementia Assessment Scale (RUDAS)
* Upper limb and trunk musculoskeletal injuries
* A score of 0 on modified Ashworth scale.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | At day one, and the end of the intervention (after 4 weeks).
  Spasticity level will be evaluated using the MAS scale. The MAS measures muscle resistance during passive stretching. The test will be applied for spastic joints of affected upper extremities. The score will be recorded as (0, 1, +1, 2, 3, 4), (0= normal tone, 4 = affected part rigid in flexion or extension). The reliability of the modified Ashworth scale is very good (kappa = .84 for interrater and .83 for intra-rater comparisons). Measurement repetition will be performed by the same assessor to avoid affecting reliability.
  The test will be conducted in the assessment quiet room, with no distractions. The participants will be supine in a treatment bed, and therapist will assess the affected upper limb spasticity once and record the result in the assessment form. The assessor will be a qualified trained occupational therapist who has worked in a clinical role treating stroke patients with hand spasticity and familiar with MAS.
Fugl-Meyer Assessment of Upper Extremity (FMA-UE) | At day one, and the end of the intervention (after 4 weeks).
  The FMA-UE looks at reflex activity, volitional movement within synergies, volitional movement mixing synergies, and volitional movement with little or no synergy. The outcome scale's 33 items are divided into four subscales: shoulder and elbow, wrist, hand, and coordination. On a three-point ordinal scale, each of these items is assessed. 2 points are granted if a movement is completely completed, 1 point is awarded if the movement is half completed, and 0 points are awarded if the movement cannot be completed.
Range of Motion Assessment | At day one, and the end of the intervention (after 4 weeks).
  The assessment of Range of Motion (ROM) for the affected upper limb in stroke patients will employ the use of a goniometer to precisely measure joint mobility across multiple planes of movement. This comprehensive evaluation entails examining the patient's ability to actively or passively articulate their affected elbow, wrist, and hand joints. The measurement of each movement will be made through the goniometer-based approach.
Numeric pain rating scale (NRS) | At day one, and the end of the intervention (after 4 weeks).
  Numeric pain scale (NRS) is an essential tool for the assessment of pain intensity. It is widely used by healthcare providers. It consists of a horizontal line where the left end is labeled "no pain" or "0," indicating the absence of pain, while the right end is labeled as "worst pain imaginable" or "10". The participants are required to mark on the line the point that shows the pain level they are experiencing. The distance from the origin of the line, which is the left end, to the participant's symbol mark is the one that is used to present a numerical value. a representation which shows pain intensity, where the higher the value the more pain there is. The NRS is taken into account as a valid and reliable scale and is usually employed in to analyze pain intensity in clinical practice and to conduct research.

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Arab Alkabeya, PhD, Study Chair — Assistant professor
Locations (1):
- Arab American University, Jenin, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tedla JS, Gular K, Reddy RS, de Sa Ferreira A, Rodrigues EC, Kakaraparthi VN, Gyer G, Sangadala DR, Qasheesh M, Kovela RK, Nambi G. Effectiveness of Constraint-Induced Movement Therapy (CIMT) on Balance and Functional Mobility in the Stroke Population: A Systematic Review and Meta-Analysis. Healthcare (Basel). 2022 Mar 8;10(3):495. doi: 10.3390/healthcare10030495. PMID 35326973
- [Background] Alashram AR, Padua E, Romagnoli C, Annino G. Effectiveness of focal muscle vibration on hemiplegic upper extremity spasticity in individuals with stroke: A systematic review. NeuroRehabilitation. 2019 Dec 18;45(4):471-481. doi: 10.3233/NRE-192863. PMID 31868686
- [Background] Alghadir AH, Anwer S, Iqbal ZA. The psychometric properties of an Arabic numeric pain rating scale for measuring osteoarthritis knee pain. Disabil Rehabil. 2016 Dec;38(24):2392-7. doi: 10.3109/09638288.2015.1129441. Epub 2016 Jan 6. PMID 26733318
- [Background] Amatya B, Khan F, La Mantia L, Demetrios M, Wade DT. Non pharmacological interventions for spasticity in multiple sclerosis. Cochrane Database Syst Rev. 2013 Feb 28;2013(2):CD009974. doi: 10.1002/14651858.CD009974.pub2. PMID 23450612
- [Background] Andringa A, van de Port I, Meijer JW. Long-term use of a static hand-wrist orthosis in chronic stroke patients: a pilot study. Stroke Res Treat. 2013;2013:546093. doi: 10.1155/2013/546093. Epub 2013 Feb 27. PMID 23533961
- [Background] Arain M, Campbell MJ, Cooper CL, Lancaster GA. What is a pilot or feasibility study? A review of current practice and editorial policy. BMC Med Res Methodol. 2010 Jul 16;10:67. doi: 10.1186/1471-2288-10-67. PMID 20637084
- [Background] Beebe JA, Lang CE. Active range of motion predicts upper extremity function 3 months after stroke. Stroke. 2009 May;40(5):1772-9. doi: 10.1161/STROKEAHA.108.536763. Epub 2009 Mar 5. PMID 19265051
- [Background] Davis EC, Barnes MP. Botulinum toxin and spasticity. J Neurol Neurosurg Psychiatry. 2000 Aug;69(2):143-7. doi: 10.1136/jnnp.69.2.143. No abstract available. PMID 10896682
- [Background] de Jong LD, Dijkstra PU, Stewart RE, Postema K. Repeated measurements of arm joint passive range of motion after stroke: interobserver reliability and sources of variation. Phys Ther. 2012 Aug;92(8):1027-35. doi: 10.2522/ptj.20110280. Epub 2012 May 10. PMID 22577062
- [Background] Eldridge SM, Lancaster GA, Campbell MJ, Thabane L, Hopewell S, Coleman CL, Bond CM. Defining Feasibility and Pilot Studies in Preparation for Randomised Controlled Trials: Development of a Conceptual Framework. PLoS One. 2016 Mar 15;11(3):e0150205. doi: 10.1371/journal.pone.0150205. eCollection 2016. PMID 26978655
- [Background] Elfil M, Negida A. Sampling methods in Clinical Research; an Educational Review. Emerg (Tehran). 2017;5(1):e52. Epub 2017 Jan 14. PMID 28286859
- [Background] Fattorini L, Ferraresi A, Rodio A, Azzena GB, Filippi GM. Motor performance changes induced by muscle vibration. Eur J Appl Physiol. 2006 Sep;98(1):79-87. doi: 10.1007/s00421-006-0250-5. Epub 2006 Aug 9. PMID 16896736
- [Background] Feigin VL, Forouzanfar MH, Krishnamurthi R, Mensah GA, Connor M, Bennett DA, Moran AE, Sacco RL, Anderson L, Truelsen T, O'Donnell M, Venketasubramanian N, Barker-Collo S, Lawes CM, Wang W, Shinohara Y, Witt E, Ezzati M, Naghavi M, Murray C; Global Burden of Diseases, Injuries, and Risk Factors Study 2010 (GBD 2010) and the GBD Stroke Experts Group. Global and regional burden of stroke during 1990-2010: findings from the Global Burden of Disease Study 2010. Lancet. 2014 Jan 18;383(9913):245-54. doi: 10.1016/s0140-6736(13)61953-4. PMID 24449944
- [Background] Francisco GE, McGuire JR. Poststroke spasticity management. Stroke. 2012 Nov;43(11):3132-6. doi: 10.1161/STROKEAHA.111.639831. Epub 2012 Sep 13. No abstract available. PMID 22984012
- [Background] Gregson JM, Leathley M, Moore AP, Sharma AK, Smith TL, Watkins CL. Reliability of the Tone Assessment Scale and the modified Ashworth scale as clinical tools for assessing poststroke spasticity. Arch Phys Med Rehabil. 1999 Sep;80(9):1013-6. doi: 10.1016/s0003-9993(99)90053-9. PMID 10489001
- [Background] Hernandez ED, Galeano CP, Barbosa NE, Forero SM, Nordin A, Sunnerhagen KS, Alt Murphy M. Intra- and inter-rater reliability of Fugl-Meyer Assessment of Upper Extremity in stroke. J Rehabil Med. 2019 Oct 4;51(9):652-659. doi: 10.2340/16501977-2590. PMID 31448807
- [Background] Katan M, Luft A. Global Burden of Stroke. Semin Neurol. 2018 Apr;38(2):208-211. doi: 10.1055/s-0038-1649503. Epub 2018 May 23. PMID 29791947
- [Background] Kerr L, Jewell VD, Jensen L. Stretching and Splinting Interventions for Poststroke Spasticity, Hand Function, and Functional Tasks: A Systematic Review. Am J Occup Ther. 2020 Sep/Oct;74(5):7405205050p1-7405205050p15. doi: 10.5014/ajot.2020.029454. PMID 32804623
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Background] Lannin NA, Herbert RD. Is hand splinting effective for adults following stroke? A systematic review and methodologic critique of published research. Clin Rehabil. 2003 Dec;17(8):807-16. doi: 10.1191/0269215503cr682oa. PMID 14682551
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Nam KE, Lim SH, Kim JS, Hong BY, Jung HY, Lee JK, Yoo SD, Pyun SB, Lee KM, Lee KJ, Kim H, Han EY, Lee KW. When does spasticity in the upper limb develop after a first stroke? A nationwide observational study on 861 stroke patients. J Clin Neurosci. 2019 Aug;66:144-148. doi: 10.1016/j.jocn.2019.04.034. Epub 2019 May 11. PMID 31088768
- [Background] Noma T, Matsumoto S, Shimodozono M, Etoh S, Kawahira K. Anti-spastic effects of the direct application of vibratory stimuli to the spastic muscles of hemiplegic limbs in post-stroke patients: a proof-of-principle study. J Rehabil Med. 2012 Apr;44(4):325-30. doi: 10.2340/16501977-0946. PMID 22402727
- [Background] Pathak A, Gyanpuri V, Dev P, Dhiman NR. The Bobath Concept (NDT) as rehabilitation in stroke patients: A systematic review. J Family Med Prim Care. 2021 Nov;10(11):3983-3990. doi: 10.4103/jfmpc.jfmpc_528_21. Epub 2021 Nov 29. PMID 35136756
- [Background] Phadke CP, Balasubramanian CK, Ismail F, Boulias C. Revisiting physiologic and psychologic triggers that increase spasticity. Am J Phys Med Rehabil. 2013 Apr;92(4):357-69. doi: 10.1097/phm.0b013e31827d68a4. PMID 23620900
- [Background] Poenaru D, Cinteza D, Petrusca I, Cioc L, Dumitrascu D. Local Application of Vibration in Motor Rehabilitation - Scientific and Practical Considerations. Maedica (Bucur). 2016 Sep;11(3):227-231. PMID 28694858
- [Background] Shiner CT, Vratsistas-Curto A, Bramah V, Faux SG, Watanabe Y. Prevalence of upper-limb spasticity and its impact on care among nursing home residents with prior stroke. Disabil Rehabil. 2020 Jul;42(15):2170-2177. doi: 10.1080/09638288.2018.1555620. Epub 2019 Mar 31. PMID 30929536
- [Background] Sommerfeld DK, Eek EU, Svensson AK, Holmqvist LW, von Arbin MH. Spasticity after stroke: its occurrence and association with motor impairments and activity limitations. Stroke. 2004 Jan;35(1):134-9. doi: 10.1161/01.STR.0000105386.05173.5E. Epub 2003 Dec 18. PMID 14684785
- [Background] Suputtitada A, Chatromyen S, Chen CPC, Simpson DM. Best Practice Guidelines for the Management of Patients with Post-Stroke Spasticity: A Modified Scoping Review. Toxins (Basel). 2024 Feb 10;16(2):98. doi: 10.3390/toxins16020098. PMID 38393176
- [Background] Suresh K, Thomas SV, Suresh G. Design, data analysis and sampling techniques for clinical research. Ann Indian Acad Neurol. 2011 Oct;14(4):287-90. doi: 10.4103/0972-2327.91951. PMID 22346019
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Welmer AK, Widen Holmqvist L, Sommerfeld DK. Location and severity of spasticity in the first 1-2 weeks and at 3 and 18 months after stroke. Eur J Neurol. 2010 May;17(5):720-5. doi: 10.1111/j.1468-1331.2009.02915.x. Epub 2009 Dec 29. PMID 20050897